CLINICAL TRIAL: NCT04054388
Title: LINE Re-education Before Colonoscopy to Confirm Optimal Bowel Cleansing: A Prospective, Colonoscopist-blinded, Randomized, Controlled Trial
Brief Title: LINE Re-education Before Colonoscopy to Confirm Optimal Bowel Cleansing
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Taipei Medical University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: 201505020
Record Dates: First submitted 2016-12-22; First posted 2019-08-13 (Actual); Last update posted 2019-08-13 (Actual); Status verified 2017-07

CONDITIONS: Bowel Cleansing
Keywords: LINE; Colonoscopy; Bowel cleansing

STUDY DESIGN:
Intervention Model Description: LINE is a popular application (App) which can share free words, photos, videos and voice messages (http://line.me/en/). LINE is available on all smart phone devices and personal computer. LINE re-education before colonoscopy to confirm optimal bowel cleansing.
Who Masked: Investigator
Masking Description: All patients will be instructed not to tell colonoscopists, nurses and investigators before, during and after the procedure about their preparation method and when they receive instructions.
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 300 Randomized to re-education group (Experimental): LINE re-education of colon preparation
  Interventions: Behavioral: LINE re-education
- 300 Randomized to control group (No Intervention): education of colon preparation 1 time in hospital

INTERVENTIONS:
Behavioral: LINE re-education
  Arms: 300 Randomized to re-education group

SUMMARY:
This is a prospective, colonoscopist-blinded, randomized, controlled study with consecutive outpatients undergoing colonoscopy in Taipei Medical University Hospital.The study would comply with the standards of the Declaration of Helsinki and current ethical guidelines. It have been approval by Taipei Medical University Institutional Review Board.

DETAILED DESCRIPTION:
Written informed consent will be obtained from all the patients. Patients will be randomized to either the LINE re-education or control group for colon preparation at the time of appointment for colonoscopy by using consecutively numbered envelopes that will contain the treatment assignments, which will be generated by a computer-allocated random digit number, in a 1:1 ratio. At least two LINE accounts for all patients or their relatives living together will be recorded in case of failure to contact. All patients will be instructed not to tell colonoscopists, nurses and investigators before, during and after the procedure about their preparation method and when they receive instructions.

ELIGIBILITY:
Inclusion Criteria:

* Outpatients aged 18-80 years undergoing colonoscopy who will provide written informed consent will be eligible for participation in the study.

Exclusion Criteria:

* history of colorectal surgery;
* severe colonic stricture or obstructing tumor;
* uncooperative mental status;
* significant ileus;
* known or suspected bowel obstruction or perforation;
* severe chronic renal failure (creatinine clearance <30 ml/min);
* severe congestive heart failure (New York Heart Association class III or IV);
* uncontrolled hypertension (systolic blood pressure >180 mm Hg, diastolic blood pressure>100 mm Hg);
* liver cirrhosis;
* toxic colitis or megacolon;
* active gastrointestinal bleeding;
* dehydration or disturbance of electrolytes;
* pregnancy or lactation; and
* hemodynamically unstable.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2015-06 (Actual); Primary Completion 2020-06 (Estimated); Study Completion 2021-06 (Estimated)

PRIMARY OUTCOMES:
Adequate bowel preparation | Day 1
  total Ottawa score <6 or Boston bowel preparation scale ≥ 6

SECONDARY OUTCOMES:
colon polyp detection rate | Day 1
  colon polyp detection rate during colonoscopy
cecal intubation rate | Day 1
  cecal intubation rate

CONTACTS AND LOCATIONS:
Overall Officials: Wei Yu Kao, M.D., Principal Investigator — Taipei Medical University Hospital
Locations (1):
- Taipei Medical University hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No